CLINICAL TRIAL: NCT05066269
Title: Normative Cardiovascular Magnetic Resonance Values for Measurement of Cardiovascular Structure and Function at MCMR
Acronym: NORMAL MCMR
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 21/WA/0272; B01254 (Other Grant/Funding Number: Manchester University NHS Foundation Trust); 299730 (Other: IRAS)
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiovascular magnetic resonance (CMR) imaging is an important clinical and research tool.

Measurements of cardiovascular structure and function can vary according to scanner vendor, scanner field strength, imaging sequence and patient population. As such, the Society for Cardiovascular Magnetic Resonance (SCMR) and the European Association for Cardiovascular Imaging (EACVI) state that local normal reference ranges for CMR measurements should be established.

This study plans to establish reference ranges for measurements of cardiovascular structure and function at the British Heart Foundation Manchester Centre for Heart and Lung Magnetic Resonance Research (MCMR). The work will underpin many other research projects and clinical practice.

The study will involve volunteers having a CMR scan that will last around 30 minutes. No contrast agent will be administered. MRI scanning uses magnetic fields to make the pictures. The NHS website describes MRI scanning as "a painless and safe procedure" and "one of the safest medical procedures available".

DETAILED DESCRIPTION:
Cardiovascular magnetic resonance (CMR) has evolved into a gold standard non-invasive imaging tool in cardiovascular medicine, especially for visualising and quantifying cardiovascular anatomy and function, and evaluating heart muscle tissue character. It has unique capabilities in the diagnostic workup of patients with suspected cardiovascular disease, and for cardiovascular research, including disease characterisation and evaluation of interventions.

Measurements of cardiovascular structure and function can vary according to MRI scanner vendor, scanner field strength, imaging sequence and local patient population. The major Societies in the field, specifically the Society for Cardiovascular Magnetic Resonance (SCMR) and the European Association for Cardiovascular Imaging (EACVI), therefore state that local normal reference ranges for CMR measurements should be established. This will be a prospective, single-centre observational study in volunteers without a history of cardiovascular disease.

The British Heart Foundation Manchester Centre for Heart and Lung Magnetic Resonance Research (MCMR), based at Manchester University NHS Foundation Trust, is a recently-opened, state-of-the-art imaging centre. Greater Manchester has the highest rates of heart disease and lung disease in England, and the highest rate of premature cardiovascular death. The overall aims of MCMR are to facilitate cardiovascular and thoracic-related research in Manchester, in order to understand why people develop heart and lung disease, diagnose heart and lung disease at an earlier stage when it is more likely to be treatable, guide patient care more effectively and evaluate new treatments, so as to improve the length, and quality of life, of people living with, or at risk of, heart and lung disease.

ELIGIBILITY:
Inclusion Criteria:

1. Written, informed consent.
2. Aged 18 and over
3. No known history of cardiovascular disease. It is recognised that it may be difficult to recruit older participants entirely free from cardiovascular disease, thus participants with relatively milder cardiovascular disease may be permitted, at the discretion of the investigator.

Exclusion Criteria:

1. Contraindication to MRI scanning, such as pacemaker, defibrillator, intraocular metal, prohibitive intracranial aneurysm clips or severe claustrophobia.
2. Unable to provide complete written or verbal consent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 healthy volunteers. separated into 12 equal sized groups. Groups will be separated by age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Normative Cardiac MRI values | 1 year
  Development of normative cardiac MRI values for MCMR unit.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Miller, Principal Investigator — University of Manchester
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
With participant consent, the pseudo-anonymised MRI scans and relevant data (such as age, sex, body surface area), may be shared with researchers in other hospitals and academic institutions. The code linking the participant number to the participant will be held at Manchester University NHS Foundation Trust and will not be shared.